CLINICAL TRIAL: NCT02836431
Title: Pharmacokinetic Study of Dexmedetomidine After Intra-nasal Dosing in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-5966
Record Dates: First submitted 2016-01-08; First posted 2016-07-19 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Heart Disease
Keywords: Pediatric; Sedation; Dexmedetomidine
MeSH Terms: conditions — Heart Diseases | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DEX 1 mcg/kg Intranasal (Experimental): Standard anesthesia care for a patient presenting for cardiac surgery includes induction of general anesthesia , placement of an endotracheal tube and an arterial line. Once these are accomplished, dexmedetomidine is administered according to group assignment.
  Interventions: Drug: Dexmedetomidine 1mcg/kg Intranasal
- DEX 2 mcg/kg Intranasal (Experimental): Standard anesthesia care for a patient presenting for cardiac surgery includes induction of general anesthesia , placement of an endotracheal tube and an arterial line. Once these are accomplished, dexmedetomidine is administered according to group assignment.
  Interventions: Drug: Dexmedetomidine 2mcg/kg Intranasal
- DEX 1 mcg/kg Intravenous (Experimental): Standard anesthesia care for a patient presenting for cardiac surgery includes induction of general anesthesia , placement of an endotracheal tube and an arterial line. Once these are accomplished, dexmedetomidine is administered according to group assignment.
  Interventions: Drug: Dexmedetomidine 1mcg Intravenous

INTERVENTIONS:
Drug: Dexmedetomidine 1mcg/kg Intranasal — DEX 1 mcg/kg Intranasal
  Arms: DEX 1 mcg/kg Intranasal
Drug: Dexmedetomidine 2mcg/kg Intranasal — DEX 2 mcg/kg Intranasal
  Arms: DEX 2 mcg/kg Intranasal
Drug: Dexmedetomidine 1mcg Intravenous — DEX 1 mcg/kg Intravenously
  Arms: DEX 1 mcg/kg Intravenous

SUMMARY:
This research study is examining the absorption of the sedative dexmedetomidine (DEX) in the blood when given by nasal spray. The study will help us determine the best dosing amount for children undergoing sedation or anesthesia with DEX.

DETAILED DESCRIPTION:
The study will be a prospective study of plasma concentrations after intranasal (1 µg/kg and 2µg/kg) and intravenous (1 µg /kg) DEX to determine the early pharmacokinetics (maximum concentration (peak) and time to peak) and bioavailability of a single intranasal dose in pediatric patients.

Dexmedetomidine sedation is commonly utilized at Cincinnati Children's Medical Center (CCHMC) and other pediatric institutions. This compound is delivered intravenously or intranasally for sedation in children with and without congenital heart disease. Intranasal DEX, though very effective for sedation, has significant variability in its onset and peak effect. Patient care will be significantly improved if factors that determine this variability in onset and peak effect can be determined. Investigators will determine the important early clinical variables of peak plasma DEX concentration (Tmax and Cmax) and the 0 - 2 hour bioavailability of intranasal DEX in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 - 48 months (inclusive) scheduled to receive anesthesia for elective cardiac surgery.
* The subject must be a candidate to receive DEX. A physician member of the Division of Cardiac Anesthesiology, not involved in the study, will make this decision.
* The subject's legally authorized representative has given written informed consent to participate in the study.

Exclusion Criteria:

* Post-natal age (PNA) < 6 months
* The subject is allergic to or has a contraindication to DEX
* Severely depressed ventricular function (ejection fraction 30% or less) on preoperative echocardiogram
* The subject has high risk cardiac conduction system disease at the discretion of the attending anesthesiologist or cardiologist.
* The subject has a hemodynamically significant coarctation or other left heart outflow obstruction
* The subject has received digoxin, beta-adrenergic antagonist, or calcium-channel antagonist on the day of the study
* The subject has received DEX within 1 week of the study date (information obtained from: parent or Medical record)
* Subject have nasal/respiratory symptoms which in the opinion of the Principal investigator, may affect intranasal drug absorption.

Ages: 6 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Maximum blood concentration level of DEX - Cmax | Blood samples will be drawn until immediately prior to Cardiopulmonary bypass, an expected average of 2 hours
  DEX concentration will be measured in the blood to determine the time point with the maximum concentration (Cmax). Blood samples will be obtained at baseline, and 10 min, 20 min, 30 min, 40 min, 50 min, 1 hour, and 2 hours after receiving DEX. If cardiopulmonary bypass (CPB) is delayed beyond two hours, one final blood sample will be obtained immediately prior to CPB.
The amount of time that a DEX is present at the maximum concentration - Tmax | Blood samples will be drawn until immediately prior to Cardiopulmonary bypass, an expected average of 2 hours
  DEX concentration will be measured in the blood to determine the time point with the maximum concentration and how long that maximum concentration lasts (Tmax). Blood samples will be obtained at baseline, and 10 min, 20 min, 30 min, 40 min, 50 min, 1 hour, and 2 hours after receiving DEX. If cardiopulmonary bypass (CPB) is delayed beyond two hours, one final blood sample will be obtained immediately prior to CPB.
Area under the curve for DEX concentration levels | Blood samples will be drawn until immediately prior to Cardiopulmonary bypass, an expected average of 2 hours
  DEX concentration will be measured in the blood samples. Blood samples will be obtained at baseline, and 10 min, 20 min, 30 min, 40 min, 50 min, 1 hour, and 2 hours after receiving DEX. If cardiopulmonary bypass (CPB) is delayed beyond two hours, one final blood sample will be obtained immediately prior to CPB.
Bioavailability of intranasal DEX relative to intravenous DEX for distribution - plasma concentration | Blood samples will be drawn until immediately prior to Cardiopulmonary bypass, an expected average of 2 hours
  Data will also be analyzed using population modeling using nonlinear mixed effect modeling (NONMEM). Investigators are limited in sampling duration to the onset time for cardiopulmonary bypass in this patient population (approximately two hours), investigators will be measuring distribution for approximately one half-life of DEX. This will allow us to estimate the important clinical parameter of relative 0-2h bioavailability of intranasal vs intravenous DEX.
Bioavailability of intranasal DEX relative to intravenous DEX for elimination - plasma concentration | Blood samples will be drawn until immediately prior to Cardiopulmonary bypass, an expected average of 2 hours
  Data will also be analyzed using population modeling using nonlinear mixed effect modeling (NONMEM). Investigators are limited in sampling duration to the onset time for cardiopulmonary bypass in this patient population (approximately two hours), investigators will be measuring elimination for approximately one half-life of DEX. This will allow us to estimate the important clinical parameter of relative 0-2h bioavailability of intranasal vs intravenous DEX.

SECONDARY OUTCOMES:
Adverse events associated with DEX administration | Participants will be followed until cardiopulmonary bypass, an expected duration of 2 hours.
  Heart rate and blood pressure are recorded by clinical staff prior to the procedure and continuously during the procedure. The heart rate and blood pressure during the time of study blood collection will be compared to the baseline vitals to determine if any adverse events occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Miller, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No